CLINICAL TRIAL: NCT01573754
Title: A Prospective Comparison of Low Dose Hydroxychloroquine and Phlebotomy in the Treatment of Porphyria Cutanea Tarda. IRB 02-435
Brief Title: Hydroxychloroquine and Phlebotomy for Treating Porphyria Cutanea Tarda
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDA-2604; R01FD002604 (FDA)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Porphyria Cutanea Tarda
Keywords: Porphyria, rare disease, orphan disease, iron metabolism
MeSH Terms: conditions — Porphyria Cutanea Tarda; Porphyrias; Rare Diseases | interventions — Hydroxychloroquine; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Low-dose hydroxychloroquine 100 mg by mouth twice weekly
  Interventions: Drug: Hydroxychloroquine
- Phlebotomy (Active Comparator): Phlebotomy 450 mL biweekly
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Drug: Hydroxychloroquine — 100 mg by mouth twice weekly
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Procedure: Phlebotomy — 450 mL every 2 weeks
  Arms: Phlebotomy

SUMMARY:
Porphyria cutanea tarda (PCT) is an iron-related disorder that responds to treatment by phlebotomy or low-dose hydroxychloroquine, but comparative data on these treatments are limited. The hypothesis is that hydroxychloroquine is noninferior to phlebotomy in terms of time to remission. Patients with well documented PCT are assigned to treatment by randomization if specific criteria are met. All patients are followed until remission - defined as achieving a normal plasma porphyrin concentration.

DETAILED DESCRIPTION:
Study Design: Pragmatic Interventional study

Primary Study Objective: To determine and compare time to remission with treatment with low-dose hydroxychloroquine or repeated phlebotomy in participants with PCT.

Secondary Study Objective(s):

1. To assess the effects of susceptibility factors on responses to treatment of PCT by these methods.
2. To determine and compare rates of recurrence of PCT after treatment with low-dose hydroxychloroquine or phlebotomy.

Study Population and Main Eligibility/ Exclusion Criteria:

Treatment:

Hydroxychloroquine 100 mg twice weekly for up to 24 months by mouth vs. phlebotomy 450 mL biweekly until target serum ferritin reached, or up to 24 months.

Safety Issues- 1. Side effects of phlebotomy or hydroxychloroquine, which are the same as in clinical practice.

Primary Outcome Measures:

1. Time to achievement of a normal plasma total porphyrin level.
2. Tolerability and safety of both treatments

Secondary Outcome Measures:

1. Time to 50% reduction in plasma porphyrin levels. 2. Time to 75% reduction in plasma porphyrin levels. 3. Time to normal urinary porphyrin levels

1. Time to disappearance of a plasma fluorescence peak at neutral pH.
2. Time to normalization of urinary total porphyrins.
3. Time to normalization of the urinary total porphyrin pattern by HPLC
4. Effects of susceptibility factors such as hepatitis C, inherited UROD deficiency, etc. on efficacy and safety of the two treatment methods.
5. Rates of recurrence after each type of treatment and the effects of susceptibility factors on recurrence rates.

Statistical Considerations (sample size and analysis plan): Time to achieving biochemical endpoints will be determined from individual subject data. Outcome measures such as time to remission will be compared using Cox proportional models to study the effects of susceptibility factors on the hazard ratio to compare the two treatments. Additional modeling will assess factors affecting the frequency of recurrence and seasonality effects using logistic regression modeling and log-rank testing, respectively.

Sponsors: National Institutes of Health (NIH)

ELIGIBILITY:
Inclusion Criteria:

* Documented porphyria cutanea tarda (PCT)
* Willing to give informed consent
* Age 18 or greater

Exclusion Criteria:

* Blistering skin lesions due to another condition

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-03-21 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl E Anderson, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Through a NIH data repository at some future time.

REFERENCES:
- [Derived] Singal AK, Kormos-Hallberg C, Lee C, Sadagoparamanujam VM, Grady JJ, Freeman DH Jr, Anderson KE. Low-dose hydroxychloroquine is as effective as phlebotomy in treatment of patients with porphyria cutanea tarda. Clin Gastroenterol Hepatol. 2012 Dec;10(12):1402-9. doi: 10.1016/j.cgh.2012.08.038. Epub 2012 Sep 14. PMID 22985607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical clinics and clinical research center
Pre-assignment Details: Diagnosis of porphyria cutanea tarda established before enrollment
Period: Overall Study
Arm/Group | Hydroxychloroquine | Phlebotomy
Started | 16 | 32
Completed | 13 | 17
Not Completed | 3 | 15
Not completed — Noncompliance or remission not achieved | 3 | 15

BASELINE CHARACTERISTICS:
Population: Gender collected, sex male and female. No race or ethnicity collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Phlebotomy | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (6.0) | 51.3 (5.0) | 50.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 5 | 15 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Remission
Description: Time to a decrease in plasma porphyrin concentration to less than 0.9 mcg/dL
Time Frame: To end of study, an average of 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Hydroxychloroquine | Phlebotomy
Number analyzed (Participants) | 13 | 17
months | 6.1 [0.9 to 10.7] | 6.9 [1.8 to 26.5]

2. Secondary Outcome: 50% Reduction in Plasma Porphyrin Level
Description: 50% reduction in plasma porphyrin level during treatment
Time Frame: To end of study, an average of 3 years
Population: Participants missed some study visits.
Measure: Median (Full Range); unit: days
Arm/Group | Hydroxychloroquine | Phlebotomy
Number analyzed (Participants) | 8 | 16
days | 44 [13 to 77] | 65 [42 to 123]

3. Secondary Outcome: 75% Reduction in Plasma Porphyrin Level
Description: Time to 75% reduction in plasma porphyrin level during treatment
Time Frame: To end of study, an average of 3 years
Population: Participants missed some study visits.
Measure: Median (Full Range); unit: days
Arm/Group | Hydroxychloroquine | Phlebotomy
Number analyzed (Participants) | 8 | 13
days | 73 [72 to 123] | 44 [40 to 238]

4. Secondary Outcome: Number of Days With Normal Urinary Porphyrin Levels
Description: Number of days to normal urinary porphyrin levels for participants treated for Porphyria Cutanea Tarda (PCT). Days are summed together for all participants for a single value in each Arm.
Time Frame: To end of study, an average of 3 years
Measure: Number; unit: days
Arm/Group | Hydroxychloroquine | Phlebotomy
Number analyzed (Participants) | 6 | 12
days | 175 | 265

ADVERSE EVENTS:
Time Frame: Up to 27 months
Arm/Group | Hydroxychloroquine | Phlebotomy
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 4/13 | 0/17
Other Adverse Events (participants affected / at risk) | 3/13 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=13) | Phlebotomy (N=17)
Death (General disorders) | 1 (1) | 0 (0) — Death from HIV/AIDS
Coronary disease (Cardiac disorders) | 2 (2) | 0 (0) — Hospitalized for coronary disease
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Hospitalized for prostate cancer surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=13) | Phlebotomy (N=17)
Suicidal thoughts (Psychiatric disorders) | 1 (1) | 0 (0) — Suicidal thoughts and hallucinations
Chest pain (General disorders) | 1 (1) | 0 (0) — Noncardiac chest pain
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Pruritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT01573754/Prot_SAP_ICF_000.pdf